CLINICAL TRIAL: NCT07177014
Title: Impact of Stress First Aid for Workers in Substance Misuse Settings
Acronym: SFA-Impact
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00008024; R61DA059887 (NIH)
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Occupational Health
Keywords: Stress First Aid; Harm Reduction Worker; Persons who use drugs; overdose prevention; community outreach workers

STUDY DESIGN:
Intervention Model Description: Cluster-randomized hybrid type I trial of SFA adapted for the harm reduction workforce (SFA/HRW) compared to a no treatment control condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Treatment (No Intervention): Control: No Treatment
- Stress First Aid for Harm Reduction Workers (Experimental): Treatment group receives Stress First Aid for Harm Reduction Workers, a 2-hour training and up to six virtual 30-minute monthly learning collaborative meetings.
  Interventions: Behavioral: Stress First Aid for Harm Reduction Workers (SFA/HRW)

INTERVENTIONS:
Behavioral: Stress First Aid for Harm Reduction Workers (SFA/HRW) — Stress First Aid for Harm Reduction Workers is a 2-hour training and up to six virtual 30-minute monthly learning collaborative meetings.
  Arms: Stress First Aid for Harm Reduction Workers

SUMMARY:
Test the effectiveness of SFA adapted for the harm reduction workforce (SFA/HRW) compared to a no treatment control condition on social-support and burnout of HRWs in a cluster-randomized hybrid type I trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Employed in a paid role as a harm reduction worker or community health/outreach worker (whose work includes harm reduction) with people who use drugs within TX, LA, AR, OK, NM and tribal areas
* Able and willing to provide informed consent

Exclusion Criteria:

- Inability to provide consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Mean Overall Burnout Assessed by the Copenhagen Burnout Inventory at 2 Months | From enrollment to 2 months after the intervention training
  A 19-item, 5-point Likert type scale, where a higher score is a worse outcome. Minimum score of 0, maximum score of 100.
Change from Baseline in the Mean Overall Social Support Assessed by the Job Content Questionnaire Social Support Sub-Scale at 2 Months | From enrollment to 2 months after the intervention training
  An 8-item; 4-point Likert-type scale, where a higher score is a better outcome. Minimum score of 8, maximum score of 40.